CLINICAL TRIAL: NCT07380269
Title: Comprehensive Follow-up and Evaluation for Cochlear Implant Patients for All Ages
Brief Title: Cochlear Implant Recipients: Comprehensive Longitudinal Evaluation
Acronym: CIRCLE
Status: Recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025192
Record Dates: First submitted 2026-01-10; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss; Hearing Loss, Sensorineural; Deafness; Cochlear Implantation; Speech Perception
Keywords: Cochlear Implant; Pediatric Cochlear Implantation; Adult Cochlear Implantation; Auditory Rehabilitation; Speech Recognition; Quality of Life; Cognitive Function; Observational Cohort
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural; Deafness | interventions — Cochlear Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cochlear Implant Recipients
  Interventions: Procedure: Cochlear Implantation

INTERVENTIONS:
Procedure: Cochlear Implantation — cochlear implantation - a surgical procedure designed to provide auditory perception to individuals with severe-to-profound sensorineural hearing loss who receive limited to no benefits from conventional amplification.

SUMMARY:
This study aims to assess hearing and speech perception, as well as quality of life, in deaf patients of all ages before and after cochlear implantation, and to explore differences across age groups and treatment subtypes, thereby providing evidence for personalized hearing and speech rehabilitation.

DETAILED DESCRIPTION:
The study aims to conduct a comprehensive evaluation of auditory and speech perception abilities, as well as overall quality of life, in patients with hearing loss across all age groups undergoing cochlear implantation. By comparing pre- and post-operative outcomes, the study will investigate how different age cohorts and subtype groups respond to cochlear implantation treatment. The findings are expected to provide critical evidence to guide the development of individualized auditory and speech rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe or greater hearing loss (≥65 dB) scheduled to receive cochlear implant (CI) treatment.
* No restrictions on age or gender.
* Native language is Mandarin Chinese.
* The subject and/or their legal guardian must provide informed consent prior to the study, voluntarily sign a written informed consent form, and be willing to undergo follow-up assessments at the specified time points.
* Ability to communicate effectively with the researcher with the help of a guardian and comply with the researcher's requirements. For young children without mature language skills, ability to cooperate with the help of a guardian.
* The subject's guardian has a correct understanding of the trial and realistic expectations of potential benefits.

Exclusion Criteria:

* Presence of other severe diseases unsuitable for cochlear implantation surgery.
* Significant psychological problems or mood disorders (e.g., notable anxiety, depression, or behavioral disorders) that would preclude cooperation with training and follow-up.
* Neurological diseases (e.g., epilepsy, cerebral palsy) that may affect auditory processing ability.
* Concurrent participation in other interventional studies involving drugs or behavioral interventions that may affect auditory rehabilitation during the study period.
* Any other condition considered by the investigator to make the subject unsuitable for participation in this clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A single-center, observational cohort of patients across all age groups (children and adults) with severe-to-profound hearing loss who are candidates for and receive cochlear implantation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Auditory Function | From enrollment until the end of the 5-year follow-up. Assessments are conducted preoperatively, at device activation, and post-activation at 4 weeks, 13 weeks, 26 weeks, 52 weeks, 2 years, 3 years, and 5 years.
  A comprehensive assessment of auditory sensitivity and daily listening abilities. Objective measures include electrophysiological tests (Auditory Brainstem Response, ABR; Auditory Steady-State Response, ASSR) for threshold estimation, particularly in non-communicative subjects. Behavioral audiometry and sound-field testing determine hearing thresholds in dB HL. Distortion Product Otoacoustic Emissions (DPOAE) assess cochlear outer hair cell function. Subjective auditory performance is evaluated using standardized questionnaires: the Categories of Auditory Performance (CAP, range 0-7, higher is better).The Parents' Evaluation of Aural/oral performance of Children (PEACH), consists of 12 core items, each rated on a 5-point scale from 0 to 4. Total scores are calculated to a percentage, ranging from 0% to 100%. A higher percent indicates better auditory and communication performance.

SECONDARY OUTCOMES:
Evaluation of Speech Function | From enrollment until the end of the 5-year follow-up. Assessments are conducted preoperatively, at device activation, and post-activation at 4 weeks, 13 weeks, 26 weeks, 52 weeks, 2 years, 3 years, and 5 years.
  Assessment of speech perception and production abilities.Objective measure of speech perception ability. The outcome is the percentage of correct responses (%) on standardized speech recognition tests, such as monosyllabic word and sentence recognition tests, administered in quiet and in noise. The score ranges from 0% to 100%. A higher percentage indicates better speech perception.Speech production ability is evaluated using the Speech Intelligibility Rating (SIR), an observer-rated scale from 1 (unintelligible) to 5 (spontaneous speech is fully intelligible).A higher rating indicates more intelligible speech.
Assessment of Psychosocial and Functional Outcomes | From enrollment until the end of the 5-year follow-up. Assessments are conducted preoperatively, at device activation, and post-activation at 4 weeks, 13 weeks, 26 weeks, 52 weeks, 2 years, 3 years, and 5 years.
  Multidimensional evaluation of the impact of cochlear implantation on cognitive status, spatial hearing, quality of life, and related symptoms. Tools include:the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE; average score, 1-5, higher=greater decline) for cognition; the Speech, Spatial and Qualities of Hearing Scale-Short Form (SSQ-12; mean item score, 0-10, higher=better) for spatial hearing; the Cochlear Implant Quality of Life (CIQoL; global score, higher=better QoL) instrument; the Vanderbilt Fatigue Scale (total score, higher=greater fatigue); and the Tinnitus Handicap Inventory (THI; total score, 0-100, higher=greater handicap).

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China